CLINICAL TRIAL: NCT02878473
Title: Liver Transplantation for the Treatment of Early Stages of Intrahepatic Cholangiocarcinoma in Cirrhotics
Brief Title: Liver Transplantation for Early Intrahepatic Cholangiocarcinoma
Acronym: LT for iCCA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-5306
Record Dates: First submitted 2016-08-17; First posted 2016-08-25 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver transplantation (Experimental): The intervention will consist of liver transplantation
  Interventions: Procedure: Deceased donor Liver Transplantation

INTERVENTIONS:
Procedure: Deceased donor Liver Transplantation — Deceased donor orthotopic liver transplantation

SUMMARY:
Diagnosis of intrahepatic cholangiocarcinoma (iCCA) is increasingly common in patients with liver cirrhosis, but these patients are denied liver transplantation (LT) by most centres due to historically poor results. Two retrospective evaluations have shown a 5 year survival ~65% in selected patients with an iCCA diagnosis at the pathology of the explanted liver. This suggests that LT can be a curative treatment if applied selectively. This study will evaluate the effectiveness of LT as a treatment for very early iCCA diagnosed in cirrhotic patients who meet the strict selection criteria. Patients with advanced cirrhosis (not candidates for resection) currently have no other curative treatment options. Participants will be allowed bridging therapies prior to receiving transplant. Participants will be followed for 5 years from the time of transplant with patient survival and disease recurrence as outcome measures.

DETAILED DESCRIPTION:
Diagnosis of intrahepatic cholangiocarcinoma (iCCA) is increasingly common in patients with liver cirrhosis. iCCA is not an indication for Liver transplantation (LT) at most transplant centres given the historically poor rates of survival and high rates of disease recurrence. A recent retrospective study shows that patients found to have very early iCCA on explant after undergoing LT for another indication, had a 5 year survival of 65% and recurrence rate of 13%.This suggests that LT can be a curative treatment if applied selectively and that it is time to reevaluate LT as a treatment option for those with very early iCCA. This study will evaluate the effectiveness of LT as a treatment for very early iCCA diagnosed in cirrhotic patients. Diagnosis of iCCA will be based upon biopsy results of a new tumor which does not present radiologically as an HCC. Patients fulfilling the strict study selection criteria will undergo a full transplant assessment and must be deemed otherwise "suitable" for liver transplant as per their centre's criteria. Patients will be treated with bridging therapies while they are on the transplant waiting list according to each center's policy. Patients with disease progression (tumor >3cm or development of extrahepatic disease) at any time prior to transplantation will be excluded. Participants will be followed for 5 years from the time of transplant with patient survival and disease recurrence as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group: 0 or 1 at all times prior to Liver Transplantation
* Absence of cancer-related symptoms
* Liver cirrhosis (any etiology)
* Patient not eligible for liver resection due to poor liver function/portal hypertension
* Biopsy proven "very early" intrahepatic cholangiocarcinoma (iCCA)
* Willing and able to provide written informed consent.
* Negative serum pregnancy test for women of childbearing potential
* Biopsy proven "very early" (single ≤2 cm) iCCa
* No vascular or biliary involvement seen in preoperative imaging
* No extra-hepatic disease seen in preoperative imaging
* Carbohydrate Antigen (CA) 19.9 values are ≤100 ng/mL

Exclusion Criteria:

* Previous or concurrent cancer (with some exceptions)
* Patients that have had previous liver resection for iCCA and the current tumor is a recurrence.
* Progression of the tumor in size >3 cm or development of extrahepatic disease.
* Large vessel invasion, defined radiologically.
* Renal dysfunction with an estimated creatinine clearance of less than 50 ml/min
* Pulmonary insufficiency
* History of cardiac disease:
* Uncontrolled infection(s)
* Known history of human immunodeficiency virus (HIV) infection.
* History of solid organ transplantation
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
5 year patient survival | 5 years

SECONDARY OUTCOMES:
disease recurrence after liver transplantation | 5 years
  5-years cumulative risk of recurrence after LT.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Sapisochin, MD, Principal Investigator — University Health Network, Toronto; Jordi Bruix, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sapisochin G, Facciuto M, Rubbia-Brandt L, Marti J, Mehta N, Yao FY, Vibert E, Cherqui D, Grant DR, Hernandez-Alejandro R, Dale CH, Cucchetti A, Pinna A, Hwang S, Lee SG, Agopian VG, Busuttil RW, Rizvi S, Heimbach JK, Montenovo M, Reyes J, Cesaretti M, Soubrane O, Reichman T, Seal J, Kim PT, Klintmalm G, Sposito C, Mazzaferro V, Dutkowski P, Clavien PA, Toso C, Majno P, Kneteman N, Saunders C, Bruix J; iCCA International Consortium. Liver transplantation for "very early" intrahepatic cholangiocarcinoma: International retrospective study supporting a prospective assessment. Hepatology. 2016 Oct;64(4):1178-88. doi: 10.1002/hep.28744. Epub 2016 Aug 24. PMID 27481548
- [Derived] Achurra P, Fernandes E, O'Kane G, Grant R, Cattral M, Sapisochin G. Liver transplantation for intrahepatic cholangiocarcinoma: who, when and how. Curr Opin Organ Transplant. 2024 Apr 1;29(2):161-171. doi: 10.1097/MOT.0000000000001136. Epub 2024 Jan 23. PMID 38258823